CLINICAL TRIAL: NCT04529564
Title: First Real-world Data on Unresectable Stage III NSCLC Patients Treated With Durvalumab After Chemoradiotherapy in Asia Area.
Brief Title: Real-world Data on Stage III NSCLC Patients Treated With Durvalumab After Chemoradiotherapy in Asia Area (PACIFIC AA)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4194R00023
Record Dates: First submitted 2020-07-01; First posted 2020-08-27 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EAP patients: The PACIFIC-AA is designed to enroll stage III unresectable NSCLC patients who received durvalumab after completion of chemoradiation therapy within an early access program in Taiwan during 2018 to 2019.

SUMMARY:
First real-world data on unresectable stage III NSCLC patients treated with durvalumab after chemoradiotherapy in Asia Area

DETAILED DESCRIPTION:
Study Design: The study is an observational review of medical records of patients diagnosed with unresectable stage III NSCLC in Taiwan, participating in an early access program (EAP). Physicians having treated patients in the EAP will be asked to recruit these patients to have their data abstracted from their medical records. Data will only be collected from routine clinical care.

Data Source(s): Centre staff will extract de-identified data from patient's medical charts. All collected data will be retrospective at time of extractions.

Study Population: Patients diagnosed with an unresectable stage III NSCLC, having not progressed after a CRT and who have received at least one dose of durvalumab following the CRT within the EAP will be the target population.

Exposure(s): Clinical characteristics, details of treatments (previous therapies, subsequent therapies), durvalumab exposure and serious AESIs Primary Outcome(s): PFS and OS. Sample Size Estimations: A target of 140 patients is estimated in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent or any locally required authorisation obtained from the patient prior to performing any protocol-related procedures
2. Adult of age ≥ 20 years at time of study entry
3. Patients must have been enrolled in one of the Pacific durvalumab EAPs

Exclusion Criteria:

1. Patients treated with durvalumab in clinical studies prior to the index date (first dose of durvalumab received within the EAP).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all patients who have participated in the EAP between 1 September 2017 until the end of EAP enrolment (5 Nov 2018 in Taiwan) and have received at least 1 dose of durvalumab prior to the present study start. Patients may participate in other clinical trials during this follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | time from initiation of the durvalumab therapy (index date) until earliest record of disease progression (estimate assessed up to 3 years)
  Defined as the time from initiation of the durvalumab therapy (index date) until earliest record of disease progression (including metastatic disease) determined by physicians' assessment, metastatic recurrence or death (if no progression) or end of follow-up (for censored observations)
Overall survival (OS) | time from durvalumab initiation date up to death or last date the patient was known to be alive (estimate assessed up to 5 years)
  Defined as the time from durvalumab initiation date up to death or last date the patient was known to be alive (for censored observations).

SECONDARY OUTCOMES:
Safety measures with retrospective collection of AESIs | time from initiation of durvalumab therapy until stop treatment (assessed up to 3 years)
  * Require concomitant use of systemic corticoids, immunosuppressants and/or endocrine therapies, or
  * Leading to durvalumab temporary interruption, or
  * Leading to durvalumab permanent discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Huggenberger, Study Director — AstraZeneca
Locations (12):
- Taiwan (12):
  - National Taiwan University Hospital-Hsinchu Branch, Hsinchu
  - Chang Gung Medical Foundation-Kaohsiung Branch, Kaohsiung City
  - Chang Gung Medical Foundation-Keelung Branch, Keelung
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194R00023&attachmentIdentifier=3e2ea266-fd3b-4a6d-91c3-2d186ff7352a&fileName=CSR-synopsis_redacted.pdf&versionIdentifier=